CLINICAL TRIAL: NCT01829347
Title: A Randomized, Open-Label, Multicenter, Controlled Study to Assess Safety and Efficacy of ELAD® in Subjects With Severe Acute Alcoholic Hepatitis (sAAH) and Lille Score Failure
Brief Title: To Assess Safety/Efficacy of ELAD in Subjects w/ Severe Acute Alcoholic Hepatitis (sAAH) and Lille Score Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to results from the VTI-208 study, the ELAD plan is being re-evaluated.
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-210
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Severe Acute Alcoholic Hepatitis
Keywords: liver failure; acute alcoholic hepatitis; patients failing steroid therapy; alcoholic hepatitis; steroid failure; Lille criteria; ELAD
MeSH Terms: conditions — Liver Failure; Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD (plus Standard of Care) (Experimental): ELAD is a human cell-based bio-artificial liver support system developed to improve survival of patients with acute liver failure and to provide liver support continuously to a subject with compromised liver function. Standard of care is predefined treatment for sAAH complications (ascites, hepatic encephalopathy, varices, etc.) per AASLD/EASL Guidelines.
  Interventions: Biological: ELAD; Other: Standard of Care treatment
- Standard of Care (Control) (Other): Standard of care is predefined treatment for sAAH complications (ascites, hepatic encephalopathy, varices, etc.) per AASLD/EASL Guidelines.
  Interventions: Other: Standard of Care treatment

INTERVENTIONS:
Biological: ELAD — ELAD is an extracorporeal system that draws blood from the subject via a dual-lumen catheter placed in a large vein, and then separates the plasma fluid (ultrafiltrate) from cellular components using a specifically-designed ultrafiltrate generator cartridge. While the cellular components are returned to the subject via the venous access, the ultrafiltrate is circulated at a high flow rate through the four metabolically-active ELAD cartridges which contain cloned, immortalized human hepatoblastoma cells (VTL C3A cells) derived from a subclone of the human hepatoblastoma cell line HepG2.
  Other Names: Human Cell-Based Bio-Artificial Liver Support System
  Arms: ELAD (plus Standard of Care)
Other: Standard of Care treatment — Standard of care treatment is predefined treatment for sAAH complications (ascites, hepatic encephalopathy, varices, etc.) per AASLD/EASL Guidelines.
  Other Names: Usual treatment for the disease

SUMMARY:
The purpose of this study is to determine if treatment with the ELAD System is safe and effective in subjects with severe acute alcoholic hepatitis and Lille score failures (Lille score >0.45).

DETAILED DESCRIPTION:
The Lille score will be used to identify subjects with an increased risk of mortality (Lille score failures). The Lille score is a prognostic model combining six reproducible variables at Day 0 and Day 7 of steroid treatment. The Lille score used in this protocol is being used independent of steroid administration during the 7 days of evaluation. A Lille score >0.45 (Lille score failure) indicates that the subject is at substantially increased risk of 30- and 90-day mortality. Subjects with severe acute alcoholic hepatitis (sAAH) are often treated with steroids as soon as their diagnosis is confirmed. This study is to assess treatment with the ELAD System in subjects who have failed per the Lille criteria, independent of steroid administration. ELAD treatment is done continuously for up to 10 days in addition to standard of care treatment. The Control group (those randomized not to receive ELAD treatment) will also get standard of care treatment. Standard of care is defined as the usual care for diet, medications, treatment of complications that may arise, etc. for sAAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 ;
* Total bilirubin ≥8 mg/dL;
* Medical history of alcohol abuse with evidence of a causal and temporal (<6 weeks) relationship to the use of alcohol and hospital admission for this episode of sAAH;
* Maddrey score ≥32
* A clinical diagnosis of severe acute alcoholic hepatitis (sAAH);
* Subject must have liver biopsy or in investigator's opinion, if risk is too great to perform liver biopsy, then clinical diagnosis is sufficient;
* Subject must be a Lille score failure (Lille score >0.45) as defined in this study.

Exclusion Criteria:

* Platelet count <50,000/mm3;
* International Normalization Ratio (INR) >3.0;
* MELD score >35;
* Evidence of infection unresponsive to antibiotics;
* Evidence of jaundice for >3 months;
* Hospital admission for any episodes of liver decompensation not related to sAAH, (other than this episode of sAAH) within the past 2 months;
* Evidence of hemodynamic instability;
* Evidence of active bleeding or of major hemorrhage defined as requiring ≥2 units of packed red blood cells to maintain a stable hemoglobin occurring within 48 hours of Screening;
* Evidence of occlusive portal vein thrombosis impairing hepatopetal flow, or evidence of bile duct obstruction;
* Evidence by physical exam, history, or laboratory evaluation of significant concomitant disease with expected life expectancy of less than 3 months;
* Clinical evidence of liver size reduction due to cirrhosis, unless Investigator interpretation of the clinical evidence indicates liver size of <10 cm or volume of <750 cc is not considered reduced for the individual subject;
* Chronic end-stage renal disease requiring chronic hemodialysis for more than 8 weeks (not classified as hepatorenal syndrome);
* Uncontrolled seizures;
* Positive serologies for viral hepatitis B or C;
* Pregnancy as determined by β-human chorionic gonadotropin (HCG) results;
* Participation in another investigational drug, biologic, or device study within one month of enrollment, except for observational studies (the observational study setting should not affect the safety and/or efficacy of the VTI-210 clinical trial);
* Currently listed or scheduled for liver transplant during the 90-day study period;
* Previous liver transplant;
* Previous participation in a clinical trial involving ELAD;
* Has a Do Not Resuscitate or a Do Not Intubate (DNR/DNI) directive (or local equivalent) or any other Advanced Directive limiting Standard of Care in place (the DNR/DNI criterion is not applicable in the UK);
* Refusal to participate in the VTI-210E follow-up study;
* Is unable to provide an address for follow-up home visits.

And other inclusion/exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stange, MD, Study Director — Vital Therapies, Inc.; Rajiv Jalan, MD, Principal Investigator — UK - Royal Free Hospital; Juan Caballeria, MD, Principal Investigator — Spain - Hospital Clinic de Barcelona; José Luis Montero, MD, Principal Investigator — Spain - Hospital Reina Sofia; Rafael Bañares, MD, Principal Investigator — Spain - Hospital Gregorio Marañon; Kalyan R Bhamidimarri, MD, Principal Investigator — FL - University of Miami Hospital; Julie Thompson, MD, Principal Investigator — MN - University of Minnesota Medical Center - Twin Cities Campus; Valentin Cuervas-Mons Martinez, MD, Principal Investigator — Spain - Hospital Universitario Puerta de Hierro - Majadahonda; Santiago Tome, MD, Principal Investigator — Spain - Hospital Clinico Universitario de Santiago de Compostela; Martín Prieto, MD, Principal Investigator — Spain - Hospital Universitario y Politécnico La Fe; Sumita Verma, MD, Principal Investigator — UK - Brighton & Sussex University Hospitals NHS Trust; Paul J Gaglio, MD, Principal Investigator — NY - Montefiore Medical Center; Manuel Romero-Gomez, MD, Principal Investigator — Spain - Hospital Universitario de Valme; Andrew deLemos, MD, Principal Investigator — NC - Carolinas Medical Center; Joanna Sayer, MD, Principal Investigator — UK - Doncaster Royal Infirmary; Lance Stein, MD, Principal Investigator — GA - Piedmont Atlanta Hospital; Javier Crespo, MD, Principal Investigator — Spain - Hospital Universitario Marques de Valdecilla; Rohit Satoskar, MD, Principal Investigator — DC - Georgetown University Hospital; David J Kramer, MD, Principal Investigator — WI - Aurora St. Luke's Medical Center; David Reich, MD, Principal Investigator — PA - Drexel University College of Medicine; Anne M Larson, MD, Principal Investigator — WA - Swedish Medical Center; Xaralambos Zervos, DO, Principal Investigator — FL - Cleveland Clinic Florida; Kirti Shetty, MD, Principal Investigator — MD - Johns Hopkins University Hospital; Simona Rossi, MD, Principal Investigator — PA - Albert Einstein Medical Center; Ram Subramanian, MD, Principal Investigator — GA - Emory University Hospital; Alexander Kuo, MD, Principal Investigator — CA - University of California San Diego; Talal Adhami, MD, Principal Investigator — OH - Cleveland Clinic Foundation; Maria Jesús Suárez, MD, Principal Investigator — Spain - Hospital Universitario de Cruces; Nikolaos T Pyrsopoulos, MD, Principal Investigator — NJ - Rutgers University Hospital; Julio Gutierrez, MD, Principal Investigator — TX - University of Texas Health Science Center, San Antonio; Andres Duarte-Rojo, MD, Principal Investigator — AR - University of Arkansas for Medical Sciences; Agustín Albillos, MD, Principal Investigator — Spain - Hospital Universitario Ramón y Cajal; Raza Malik, MD, Principal Investigator — MA - Beth Israel Deaconess Medical Center; Markus Busch, MD, Principal Investigator — Germany - Medizinische Hochschule Hannover; Anupama Duddempudi, MD, Principal Investigator — NY - North Shore University Hospital; Marco Antonio Olivera-Martinez, MD, Principal Investigator — NE - University of Nebraska Medical Center; Eckart Schott, MD, Principal Investigator — Germany - Charité Campus Virchow-Klinikum Medizinische Klinik
Locations (39):
- United States (21):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, San Diego, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Hospital, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Johns Hopkins University Hospital, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center - Twin Cities Campus, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers University Hospital, Newark, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Germany (2):
  - Charité Campus Virchow-Klinikum Medizinische Klinik, Berlin
  - Medizinische Hochschule Hannover, Hanover
- Spain (10):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (6):
  - Barts Health NHS Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Royal Free Hospital, Hampstead, London
  - NHS Tayside, Dundee, Scotland
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire
  - Brighton & Sussex University Hospitals NHS Trust, Brighton

REFERENCES:
- [Derived] Pares A, Mas A. Extracorporeal liver support in severe alcoholic hepatitis. World J Gastroenterol. 2014 Jul 7;20(25):8011-7. doi: 10.3748/wjg.v20.i25.8011. PMID 25009371
- See also: Sponsor's website — http://www.vitaltherapies.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ELAD (Plus Standard of Care): Participants randomized to the ELAD group received ELAD treatment plus protocol-directed Standard of Care treatment for a period of up to 10 days, followed by Standard of Care treatment through Study Day 91.
- Standard of Care (Control): Participants randomized to the Control group received protocol-directed Standard of Care treatment in accord with AASLD and EASL guidelines for up to 91 days.
Period: VTI-210
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control)
Started | 9 | 9
Completed | 3 | 6
Not Completed | 6 | 3
Not completed — Death | 5 | 3
Not completed — Withdrawal by Subject | 1 | 0
Period: VTI-210E
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control)
Started | 3 | 6
Completed | 0 | 0
Not Completed | 3 | 6
Not completed — Death | 2 | 1
Not completed — Study terminated prematurely | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (7.29) | 50.0 (9.79) | 48.1 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 1 | 5
  United Kingdom | 2 | 2 | 4
  Spain | 3 | 6 | 9
Baseline MELD Score [Mean (Standard Deviation); unit: MELD Score] — The Model for End-stage Liver Disease (MELD) score is calculated by the following formula: MELD SCORE= 0.95 x LOGc (creatinine g/dL) + 0.378 x Logc (bilirubin mg/dL) + 1.120 x Logc (INR) + 0.643. The 3 tests, bilirubin (liver function), INR (blood clotting), and creatinine (kidney function), can all be affected by advanced liver disease. The scores range from 6 in a healthy person to 40. A person with a MELD score of 40 might very well be quite ill and in a hospital intensive care unit. A higher baseline MELD score value represents a worse outcome. This study excluded patients with a MELD >35.
  MELD Score | 27.531 (2.8870) | 26.323 (2.8524) | 26.962 (2.8484)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary endpoint of the study was a comparison of overall survival (OS) between ELAD-treated and Control groups, with protocol VTI-210E providing additional survival data up to a maximum of 5 years, that was included as available at the time of database lock (11 July 2016).
Time Frame: Up to at least Study Day 91, with protocol VTI-208E providing additional survival data at the time of database lock (11 July 2016), approximately 27 months
Measure: Count of Participants; unit: Participants
Groups:
- ELAD (Plus Standard of Care): Participants randomized to the ELAD group received ELAD treatment plus protocol-directed standard of care treatment for a period of up to 10 days followed by standard of care treatment through Study Day 91.
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control)
Number analyzed (Participants) | 9 | 9
Participants | 2 | 5
Statistical Analysis 1: Comparison: ELAD (Plus Standard of Care) vs Standard of Care (Control); The primary endpoint was assessed using a Kaplan-Meier survival analysis of the Intent-to-Treat (ITT) population utilizing a log-rank test; Test type: Superiority; p = 0.076, Log Rank; Hazard Ratio (HR) = 0.310, 95% CI 2-sided [0.085 to 1.133]

2. Secondary Outcome: Proportion of Survivors at Study Day 91.
Description: Assess the proportion of survivors at Study Day 91.
Time Frame: Up to Study Day 91.
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control)
Number analyzed (Participants) | 9 | 9
Participants | 5 | 6
Statistical Analysis 1: Comparison: ELAD (Plus Standard of Care) vs Standard of Care (Control); Test type: Superiority; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Time Frame: Randomization through Study Day 91.
Description: Additional relevant information: It should be noted that the outcome of the serious adverse events is recorded as the subject status at Study Day 91. Note, one serious adverse event (melaena) was ongoing at Study Day 91, and ultimately resulted in death of the subject at Study Day 91, at which time the subject had entered VTI-210E.
Arm/Group | ELAD (Plus Standard of Care) | Standard of Care (Control)
All-Cause Mortality (participants affected / at risk) | 7/9 | 4/9
Serious Adverse Events (participants affected / at risk) | 6/9 | 5/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD (Plus Standard of Care) (N=9) | Standard of Care (Control) (N=9)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD (Plus Standard of Care) (N=9) | Standard of Care (Control) (N=9)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (4) | 4 (4)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 3 (3) | 0 (0)
Medical device complication (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (6) | 2 (3)
Xerosis (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (7) | 2 (4)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (2) | 0 (0)
Vulval cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fluid overall (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Critical illness myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asterixis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (4) | 1 (1)
Irregular sleep phase (Nervous system disorders) | 0 (0) | 1 (1)
Stupor (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Flat affect (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (7) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early after enrollment of only 18 out of 150 planned subjects due to findings from previous VTI-208 study. Thus, sample size of VTI-210 was very small leading to statistical analyses that cannot be meaningfully interpreted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes